CLINICAL TRIAL: NCT00858572
Title: A Phase 1 Study of the HSP90 Inhibitor, STA-9090, Administered Twice Weekly in Subjects With Hematologic Malignancies
Brief Title: STA-9090 for Treatment of AML, CML, MDS and Myeloproliferative Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9090-03
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: AML; CML; MDS; Myeloproliferative Disorders
Keywords: Synta; STA-9090; AML; CML; MDS; myeloproliferative disorder; hematologic malignancy; ganetespib
MeSH Terms: conditions — Myeloproliferative Disorders; Hematologic Neoplasms | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental)
  Interventions: Drug: STA-9090 (ganetespib)

INTERVENTIONS:
Drug: STA-9090 (ganetespib) — Chemotherapy agent

SUMMARY:
The purpose of this study is to characterize the safety and efficacy of STA-9090 (ganetespib) in subjects with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria

* Males and females 18 years or older
* Eligible subjects must have one of the following relapsed or refractory hematologic malignancies: AML, MDS, CML, or myeloproliferative disorders as defined in the protocol
* Must have acceptable organ function during screening as defined in the protocol

Exclusion Criteria

* Pregnant or breast-feeding women
* Patients must meet the washout periods for prior chemotherapies and radiation
* History of stroke within 6 months of treatment
* Poor venous access for study drug administration
* Treatment with chronic immunosuppressants
* Other severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of STA-9090 (ganetespib) in subjects with hematologic malignancies | Feb 2011
To assess preliminary evidence of anti-neoplastic activity | Feb 2011
To assess the pharmacokinetics of STA-9090 (ganetespib) when administered as a short-term intravenous infusion | Feb 2011

SECONDARY OUTCOMES:
To assess changes in biomarkers following study drug administration | Feb 2011
To investigate drug exposure levels/plasma concentrations and correlations with efficacy and safety parameters | Feb 2011
To assess the impact of variations in drug metabolizing enzymes (DME pharmacogenomics) on the pharmacokinetics of STA-9090 (ganetespib) | Feb 2011

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Boston, Massachusetts
  - New York, New York
  - San Antonio, Texas